CLINICAL TRIAL: NCT03692299
Title: Efectividad de Saccharomyces Oulardii Para Reducir Los síntomas Gastrointestinales y Evitar el Sobrecrecimiento Bacteriano en Esclerosis sistémica
Brief Title: Effectiveness of Saccharomyces Boulardii for Gastrointestinal Bacterial-overgrowth in Systemic Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Maria del Pilar Cruz Dominguez, Chief of Researh Division, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2015-3501-72
Record Dates: First submitted 2016-12-20; First posted 2018-10-02 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Systemic Sclerosis; Small Intestinal Bacterial Overgrowth
Keywords: Systemic Sclerosis; Small Intestinal Bacterial Overgrowth; Saccaromyces boulardii
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Open Clinical Trial
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saccaromyces boulardii oral tablet (Active Comparator): Saccharomyces boulardii Oral Tablet 200 mg b.i.d. during 2 weeks, followed by a 2-week rest period and then again 200 mg b.i.d. during 2 consecutive months.
  Interventions: Drug: Saccharomyces Boulardii Oral Tablet
- Metronidazole plus S. boulardii (Active Comparator): Metronidazole 500 mg b.i.d during 1 week, followed by a 3-week rest period and then again 500 mg b.i.d during 2 consecutive months.
  Interventions: Drug: Saccharomyces Boulardii Oral Tablet; Drug: Metronidazole
- Metronidazole (Active Comparator): Metronidazole 500 mg b.i.d during 1 week, plus Saccharomyces boulardii 200 mg b.i.d. during 1 week, follow for only Saccharomyces 200 mg b.i.d. for one another week, 2-week rest period and then this regimen is repeated for two consecutive months.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Saccharomyces Boulardii Oral Tablet — Saccharomyces boulardii 200 mg b.i.d. during 2 weeks, followed by a 2-week rest period and then again 200 mg b.i.d. during 2 consecutive months.
  Other Names: Saccaromyces boulardii
  Arms: Metronidazole plus S. boulardii; Saccaromyces boulardii oral tablet
Drug: Metronidazole — Metronidazole 500 mg b.i.d during 1 week, followed by a 3-week rest period and then again 500 mg b.i.d during 2 consecutive months
  Other Names: Metronidazole alone
  Arms: Metronidazole; Metronidazole plus S. boulardii

SUMMARY:
Introduction. Autonomic dysfunction, smooth muscle fibrosis and vascular damage lead to small intestinal bacterial overgrowth (SIBO) in Systemic Sclerosis (SSc). SIBO is characterized by diarrhea, abdominal pain, bloating, malabsorption and malnutrition.

Aim. To evaluate the efficacy and safety of Saccharomyces boulardii in combination with metronidazole for 2 months for reducing gastrointestinal symptoms (NIH-PROMIS) and preventing bacterial overgrowth (hydrogen breath test) versus the standard treatment in patients with systemic sclerosis.

Method. Controlled clinical trial conduct in patients with SSc (ACR-EULAR 2015) who signed informed consent. NIH PROMIS®questionarie will be apply to evaluate gastrointestinal symptoms and classify in not symptomatic, least, mildy, moderately and most symptomatic. Glucose HBT will be apply after 14 hours fast, oral hygiene and 30 days free of antibiotics to evaluate SIBO. Patients with negative HBT and symptoms associated to glucose ingestion will repeat test with lactulose. Patients will be aleatorized into 1. Saccharomyces boulardii, 2. Metronidazole and 3. Metronidazole plus Saccharomyces boulardii.

All data will be analyzed using SPSS software. It will be used parametric statistics for normally distributed variables and nonparametric statistics for free distribution.

DETAILED DESCRIPTION:
The study will be carried out with prior authorization from the Local Research and Ethics Committee. Patients entitled to our healthcare services and complying with screening criteria will be included.

Patients with scleroderma included in our database will be invited to participate in the study through a telephone call. Patients complying with the screening criteria and accepting to participate in the study will be given a date for an interview.

On the day of the interview, they will be given the informed consent form. Once it has been signed, they will be asked to complete the NIH PROMIS questionnaire for gastrointestinal symptoms. In order to validate the questionnaire, it will be translated from English into Spanish, then back-translated from Spanish into English and submitted to a panel of gastroenterology experts. Once patients have completed the questionnaire, a Cronbach's alpha test will be carried out. Another visit will be scheduled two weeks later to perform the hydrogen breath test and patients will be given instructions to help them complete the test.

On the second visit (two weeks later), the following parameters will be recorded: weight (measured with a Seca scale without shoes and wearing a hospital gown), height, abdominal girth at the level of the navel (using a measuring tape), and patients will take the hydrogen breath test (Gastrolyzer instrument). Patients with a positive result will be randomly assigned to one of three groups: group 1 (Saccharomyces boulardii), group 2 (metronidazole) or group 3 (metronidazole + Saccharomyces boulardii).

Group 1. Saccharomyces boulardii 200 mg b.i.d. during 2 weeks, followed by a 2-week rest period and then again 200 mg b.i.d. during 2 consecutive months.

Group 2. Metronidazole 500 mg b.i.d during 1 week, followed by a 3-week rest period and then again 500 mg b.i.d during 2 consecutive months.

Group 3. Metronidazole 500 mg b.i.d during 1 week, plus Saccharomyces boulardii 200 mg b.i.d. during 1 week, follow for only Saccharomyces 200 mg b.i.d. for one another week, 2-week rest period and then this regimen is repeated for two consecutive months.

Each group will be given written instructions regarding the drug use. At the end of the first cycle, another visit will be scheduled to check for treatment compliance (remaining capsules will be counted) and patients will be given a new drug supply for the following month. Participants will also be asked to complete a form recording GI symptoms and potential adverse events. At the end of each treatment cycle, patients will have to take the hydrogen breath test, to complete the NIH PROMIS questionnaire and their weight and height will be measured. At the end of the second cycle, the statistical analysis will be carried out.

If the episodes of diarrhea or abdominal distension persist for more than 2 weeks, the probiotic treatment will be withdrawn and the patient will be given the standard treatment.

- NIH-PROMIS questionnaire

This questionnaire is used to evaluate gastrointestinal symptoms through 60 questions divided into 8 domains:

1. Heartburn / reflux (13 items)
2. Disrupted swallowing (7 items)
3. Diarrhea (5 items)
4. Fecal incontinence (4 items)
5. Nausea / vomiting (4 items)
6. Constipation (9 items)
7. Belly pain (6 items)
8. Gas / bloating (12 items)

Each question has 5 possible answers scored from 1 to 5. The physician will give the questionnaire to the patient and will cross out the answer corresponding to symptoms' severity. At the end of each domain, individual scores are added to calculate a raw score, from which a percentile is obtained. This finally leads to a symptom severity score.

- Hydrogen breath test

The patient should prepare for the test by following the instructions from Appendix 3. On the day of the test, the patient will blow into the mouthpiece of the breath hydrogen monitor after taking a deep breath. First, a baseline sample will be taken. The hydrogen baseline level must be under 10 ppm. A baseline hydrogen content over 10 ppm strongly suggests bacterial overgrowth. Then, the patient has to ingest, within 3 to 5 minutes, 50 g of glucose dissolved in 250 ml of water. Samples of exhaled air (alveolar air) will be taken after 15, 30, 45, 60, 90, 120 and 150 minutes from the moment the patient has finished taking all the glucose. Patients with values under 10 ppm but having symptoms associated to glucose ingestion (headache, dizziness, nausea, vomiting, distension, hyperperistalsis, tiredness) will have to take the test again using 50 g of lactulose dissolved into 250 ml of water.

In presence of bacterial overgrowth, carbohydrates used as substrate (glucose or lactulose) typically produce two peaks: an early increase of 10 ppm is observed when the substrate comes into contact with small intestinal bacteria, and then, after one hour, a second peak (a lot larger than the first one) is observed, being produced by normal colonic flora fermenting the remaining substrate The two peaks may merge and form an early plateau. The test is positive for bacterial overgrowth if the hydrogen level exceeds 10 ppm within 30 minutes of the lactulose dose or if baseline hydrogen levels exceed 20 ppm. If there is no response to the substrate, a flat curve can be observed and it should be interpreted as an impairment of the gut by antimicrobial agents prior to the test, pH changes in the feces at colon level, extremely slow intestinal transit and predominance of methane-producing bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Social security beneficiaries affiliated to the "LA RAZA" UMAE HECMN
* Adults over 18 years old
* Male or female subjects
* Diagnosed with scleroderma (2013 ACR-EULAR)
* Score above the 25th percentile in NIH-PROMIS questionnaire
* Positive result (> 10 ppm) in the hydrogen breath test
* Normal leukocyte and lymphocyte profiles
* Patients who accept to participate in the study by signing the informed consent form

Exclusion Criteria:

* Gastrointestinal diseases already diagnosed and not associated to systemic sclerosis
* Comorbidities associated to visceral diseases (diabetes, amyloidosis or other infiltrative diseases)
* Currently under biological treatment (or history of biological treatment in the last year) with cyclophosphamide and > 10 mg prednisone or equivalent
* Allergy or contra-indications to metronidazole or to Saccharomyces boulardii,
* Central venous catheter carriers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-06; Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Small intestinal Bacterial Overgrowth (Presence or absence) | baseline, second month
  Small intestinal Bacterial Overgrowth will be measured by a breath test using a hydrogen monitor. Hydrogen is part of the bacteria metabolism and can be detected in breath. it can be quantified in parts per million. We wil consider presence of Small intestinal Bacterial Overgrowth if a measure > 10 part per million is obtained in our patients. We will compare the presence or abscense of Small intestinal bacterial overgrowth after the intervention.

SECONDARY OUTCOMES:
Intensity of gastrointestinal symptoms | baseline, second month
  The patients that will be included in our protocol are characterized by having important gastrointestinal symptoms, inherent to its disease. The NIH Patient-Reported Outcomes Measurement Information System (NIH-PROMIS) is a tool used to assess gastrointestinal symptoms. It consist on a 48 items survey that can be answered in less than 15 minutes. A percentile is obtained after collecting data from each survey, and accordingly, we can classify the intensity of gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pilar Cruz-Domínguez, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Maria del Pilar Cruz Dominguez, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Collinot G, Madrigal-Santillan EO, Martinez-Bencomo MA, Carranza-Muleiro RA, Jara LJ, Vera-Lastra O, Montes-Cortes DH, Medina G, Cruz-Dominguez MP. Effectiveness of Saccharomyces boulardii and Metronidazole for Small Intestinal Bacterial Overgrowth in Systemic Sclerosis. Dig Dis Sci. 2020 Apr;65(4):1134-1143. doi: 10.1007/s10620-019-05830-0. Epub 2019 Sep 23. PMID 31549334